CLINICAL TRIAL: NCT06836713
Title: Surgical Risk Stratification As an Instrument for Innovation in Cardiac Surgery Programs in the Unified Health System of the São Paulo State
Brief Title: Paulista Cardiovascular Surgery Registry I
Acronym: REPLICCAR I
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: 385312109
Record Dates: First submitted 2022-04-28; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2022-04

CONDITIONS: Health Sciences; Medicine; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgical Risk Stratification — Database implementation to formulate a regional risk score

SUMMARY:
Cardiovascular diseases represent the greatest burden of morbidity and mortality for the health system and cardiac surgery has an important impact on their resolutivity. The association and correlation of patients' demographic and clinical relevant information with the resources required for each stratum represent the possibility to adapt, improve and innovate into the healthcare programs. This project aims to remodel the "InsCor" risk score for the formulation of the SP- SCORE (Sao Paulo System for Cardiac Operative Risk Evaluation) in order to better reflects the complexity of cardiac surgical care, The participating hospitals include the Health Technology Assessment Centers in of the Health Secretarlat'HTA Network of São Paulo State (HTA-NATSs / SES-SP). The SP-SCORE will use 10 variables of the InsCor model and others 8 variables with presumed influence in Brazil. The primary endpoints are morbidity and mortality. This project will contribute for the SUS- SP regionalized health-care (RRAS) sustainability and financing of the CABG and/or heart valve surgery programs promoting equitable allocation, increasing access and effectiveness, as well as characterizing the magnitude of available resources and its impact. (AU)

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent isolated coronary artery bypass grafting (CABG) surgery, mitral valve surgery, aortic valve surgery, combined mitral + aortic valve surgery, and CABG + heart valve surgery

Exclusion Criteria:

* Patients operated on in an emergency or rescue situation and who underwent percutaneous or transcatheter procedures were excluded from this analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery (coronary artery bypass grafting and/or heart valve surgery)
Sampling Method: Non-Probability Sample
Enrollment: 5222 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | Mortality until 30 days after the susrgical procedure
  Mortality until 30 days after the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Augusto F Lisboa, PhD, Study Director — instituto do Coração, Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de SaoPaulo, Sao Paulo, SP, BR; Nakazone, Principal Investigator

IPD SHARING:
Plan to Share IPD: No
The data underlying this study cannot be made available due to ethical restrictions; patients did not consent to their de-identified data being publicly shared. De-identified data can be made available to qualified researchers under their responsibility and assuming the penalties if public disclosure of the data. Data requests should be sent to Renata do Val, Director of the Scientific Committee, Ethics Committee of the Heart Institute-University of São Paulo (renata.doval@incor.usp.br, http://www.incor.usp.br/sites/incor2013/index.php/equipe/16-pesquisa/comissao-cientifica/158-fale-conosco) or Prof. Dr. Alfredo José Mansur, Coordinator, Comissão de Ética para Análise de Projetos de Pesquisa-CAPPesq (cappesq.adm@hc.fm.usp.br, http://www.hc.fm.usp.br/index.php?option=com_content&view=article&id=243:comissao-de-etica-para-analise-de-projetos-de-pesquisa-do-hcfmusp&catid=23&Itemid=229).